CLINICAL TRIAL: NCT03224962
Title: Reliability of Fluorescent Camera and Caries Detection Dye Versus Visual- Assessment in Diagnosis of Occlusal Carious Lesion in Adult Patients: Invivo Diagnostic Study
Brief Title: Reliability of Fluorescent Camera in Diagnosis of Occlusal Carious Lesion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Maher Zenhom Abd El Rahman, Assistant lecturer, Cairo University
Other Study IDs: CEBC-CU-2017-07-28
Record Dates: First submitted 2017-07-13; First posted 2017-07-21 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Caries
Keywords: pit and fissure caries
MeSH Terms: conditions — Van der Woude syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diagnostic tool: Light induced fluorescence camera Caries detection dye. visual assessment method (ICDAS criteria)
  Interventions: Device: fluorescence camera

INTERVENTIONS:
Device: fluorescence camera — drug - diagnostic test
  Other Names: Caries detection dye.; visual assessment method (ICDAS criteria)

SUMMARY:
This study will be conducted to compare the diagnostic predictive values of a light induced fluorescence camera and Caries detection dye versus visual assessment method in identification of occlusal carious lesion.

DETAILED DESCRIPTION:
A total of 43 volunteer patients will be assigned in this study. Each patient must have at least two occlusal carious lesions. Each lesion will be evaluated by three diagnostic methods (D), where D1 represents light induced fluorescence camera, D2 represents Caries detection dye. And D3 represents visual assessment method (ICDAS criteria)

ELIGIBILITY:
Inclusion Criteria:

* Patients should be over 18 Years old
* Patient should have good oral hygiene and general health
* patients With at least 2 non-cavitated first and/or second molar teeth in each quadrant of maxilla or mandible

Exclusion Criteria:

* Known allergy to any component of the dyes used.
* Patients having caries at proximal, buccal, lingual surface.
* Previously placed sealants or restorations.
* Bruxism or malocclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult populations suffering from occlusal caries.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Reliability and level of agreement between operators for all diagnostic methods. | 3 months
  It will be assessed using reliability & reproducibility by kappa strength measuring unit

CONTACTS AND LOCATIONS:
Overall Officials: Mona I Riad, Professor, Principal Investigator — Conservative Dentistry Department, Faculty of Oral and Dental Medicine, Cairo University, Egypt.

IPD SHARING:
Plan to Share IPD: Undecided